CLINICAL TRIAL: NCT00114699
Title: A Phase 1, Randomized, Placebo-Controlled, Single-Injection, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ccr5mab004 (Human Monoclonal Igg4 Antibody To Ccr5) in Hiv-1 Seropositive Individuals Who Are Not Receiving Concurrent Antiretroviral Therapy
Brief Title: Safety and Efficacy of an Antibody to CCR5 in Individuals With HIV Who Are Not Currently on Antiretroviral Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CCR5-HV01
Record Dates: First submitted 2005-06-16; First posted 2005-06-17 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: CCR5mAb004

SUMMARY:
This is a phase 1, randomized, placebo-controlled, dose-escalation study of CCR5mAb004 in HIV-1 seropositive individuals who are not receiving concurrent antiretroviral therapy. Subjects will be randomly assigned to receive a single intravenous (IV) infusion of one of four dose levels of CCR5mAb004 or matching placebo. A minimum of 10 subjects will be randomized to each cohort at a ratio of 4:1 (active:placebo). A minimum of 40 and maximum of 60 subjects will be enrolled. This study will be conducted at up to 10 sites in the United States.

Subjects in each cohort will be followed for 56 days after study agent administration. The safety, tolerability, and immunogenicity of CCR5mAb004 will be evaluated based on physical examination, adverse event (AE) reporting, and clinical laboratory tests. Blood will be collected at specified times for the determination of CCR5mAb004 serum concentrations, HIV-1 RNA levels, and CD4+ and CD8+ cell counts. If CD4+ cell counts are less than 200 during the study period, the subject should be offered standard-of-care per HIV treatment guidelines that may include the initiation of appropriate anti-retroviral therapy (AVR). CCR5mAb004 pharmacokinetic (PK) and pharmacodynamics (PD) will be measured over the 56-day study period. Anti-CCR5mAb004 antibody titers will be assessed prior to dosing on Day 0 and on Day 28 and Day 56.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection confirmed by enzyme immunoassay (EIA) and Western blot.
* Age 18 to 64 years.
* HIV-1 RNA > 5000 copies/mL.
* CD4+ T cell count > 250 cells/uL.
* Treatment naïve, or off antiretroviral treatment for at least 30 days prior to screening and 60 days prior to Day 0
* CCR5 tropism confirmed by R5 PhenoSense assays.

Exclusion Criteria:

* CXCR4 tropic or dual tropic virus at screening.
* Laboratory values of Grade 3 or greater according to the Modified Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Tables.
* History of Category C AIDS-defining illness according to the 1993 Centers for Disease Control and Prevention (CDC) AIDS surveillance definition.
* History of any medical disease or condition that makes the subject (in the opinion of the investigator) unsuitable for the study.
* Malignancy within the past 5 years (except for basal carcinomas of the skin and in situ cancers of the cervix).
* Females who are pregnant or breastfeeding, or who plan to become pregnant during the study.
* Subjects whose dosage or number of prescription medications has changed within 30 days prior to screening
* Positive for hepatitis B surface antigen (HBsAg) or antibody to hepatitis C virus (HCV).
* Positive alcohol or drug screen

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-04; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The major safety endpoints are AE rates and laboratory abnormalities through Day 56.

SECONDARY OUTCOMES:
The efficacy endpoints include change from baseline HIV-1 RNA levels (including viral kinetics) through Day 56, and change from baseline CD4+ and CD8+ cell counts through Day 56.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - AIDS Research Alliance, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Fort Lauderdale, Florida
  - The Orlando Immunology Center, Orlando, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University Hospitals of Cleveland, Cleveland, Ohio
  - OSU Medical Center, Columbus, Ohio